CLINICAL TRIAL: NCT00092170
Title: A Prospective, Multicenter, Randomized, Open-Label, Comparative Study to Evaluate the Safety, Tolerability, and Efficacy of Ertapenem Sodium ( MK0826) Versus Ticarcillin/Clavulanate in the Treatment of Hospital-Acquired Pneumonia, Complicated Intra-Abdominal Infections, and Acute Pelvic Infections in Pediatric Patients
Brief Title: An Investigational Agent for the Treatment of Complicated Intra-Abdominal Infections or Acute Pelvic Infections (0826-038)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 0826-038; 2004_062
Record Dates: First submitted 2004-09-21; First posted 2004-09-24 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Infections; Pelvic Infections
Keywords: Intra-abdominal infections; Acute pelvic infections
MeSH Terms: conditions — Infections; Pelvic Infection; Intraabdominal Infections | interventions — Ertapenem; Clavulanic Acid

INTERVENTIONS:
Drug: MK0826, ertapenem sodium
Drug: Comparator: Ticarcillin/Clavulanate

SUMMARY:
The purpose of this study is to determine the effect of an approved medication for adults for an investigational use in pediatric patients 3 months to 17 years for the treatment of complicated intra-abdominal infections or acute pelvic infections.

DETAILED DESCRIPTION:
The duration of treatment is 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 3 months to 17 years with intra-abdominal infection or acute pelvic infection

Exclusion Criteria:

* Immune problems
* Kidney problems

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100
Dates: Start 2002-03; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Efficacy response at post treatment follow up assessment. Clinical and/or laboratory drug-related SAEs during study drug therapy plus 14 days post therapy

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Yellin AE, Johnson J, Higareda I, Congeni BL, Arrieta AC, Fernsler D, West J, Gesser R. Ertapenem or ticarcillin/clavulanate for the treatment of intra-abdominal infections or acute pelvic infections in pediatric patients. Am J Surg. 2007 Sep;194(3):367-74. doi: 10.1016/j.amjsurg.2007.01.023. PMID 17693284
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html